CLINICAL TRIAL: NCT03186859
Title: Effects of Dietary Intervention and Surgery on NAFLD (Non-Alcoholic Fatty Liver Disease)
Acronym: EDISON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 219190
Record Dates: First submitted 2017-05-23; First posted 2017-06-14 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2020-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non Alcoholic Fatty Liver; Bariatric Surgery Candidate; Obesity, Morbid
Keywords: non-alcoholic fatty liver disease; bariatric surgery
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity, Morbid | interventions — Gastric Bypass; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roux-en-Y Gastric Bypass (RYGB) surgery (Active Comparator)
  Interventions: Procedure: Roux-en-Y Gastric Bypass (RYGB) surgery
- Sleeve Gastrectomy (SG) surgery (Active Comparator)
  Interventions: Procedure: Sleeve Gastrectomy (SG) surgery

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass (RYGB) surgery — RYGB operation using surgeons' standard technique
  Arms: Roux-en-Y Gastric Bypass (RYGB) surgery
Procedure: Sleeve Gastrectomy (SG) surgery — SG surgery using surgeons' standard technique
  Arms: Sleeve Gastrectomy (SG) surgery

SUMMARY:
Approximately 90% of people undergoing bariatric surgery have NAFLD, which is a condition where fat accumulates in the liver and can lead to inflammation and scarring. It mostly causes no symptoms, however, in the most advanced cases there is an increased risk of liver cancer or liver failure.

NAFLD is currently managed by weight loss and treating associated diseases such as diabetes. No medicines have been licensed to directly treat it but bariatric surgery has been shown to be usually beneficial, although it is unknown whether some operations are better than others. It is also unclear whether this is due to general weight loss or other factors.

This study will be conducted in a hospital setting and aims to determine what changes in liver fat and fat processing occur after pre-operative low calorie diet and the two most common types of bariatric surgery (Roux-en-Y Gastric Bypass and Sleeve Gastrectomy.

Participants will have ten study visits, four of which may be combined with NHS appointments. Participants will undergo investigations including MRI scans to measure changes in NAFLD and DEXA scans to measure changes in fat and fat-free mass (FFM). Participants will also undergo mixed meal testing to which stable isotopes (deuterated water and 13c-palmitate) will be added to allow changes in fat processing to be detected. In addition to samples taken as part of NHS care, blood, urine, liver and fat (visceral and subcutaneous (abdominal and gluteal)) will be used for research. Visits will take place before and after low calorie diet and bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Bariatric surgery is already planned for the participant
* Participant is willing and able to give informed consent for participation in the study.
* Aged ≥18 or ≤75 years.
* Body Mass Index ≥35 ≤55 kg/m2

Exclusion Criteria:

* Contraindication to MRI
* Prior or current participation in a CTIMP that could affect study results
* History of alcoholism or a greater than recommended weekly alcohol intake (14 units per week)
* History of albumin allergy
* Anticoagulant treatment
* Pregnant or nursing mothers
* Type 2 Diabetes
* A liver disease other than NAFLD
* Histological confirmation of lack of NAFLD on liver biopsy
* Large hiatus hernia (that would prohibit Sleeve Gastrectomy)
* Active gastrooesophageal reflux disease (that would prohibit Sleeve Gastrectomy)
* Active malabsorptive intestinal disease (that would prohibit Roux-en-Y Gastric Bypass surgery)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Change in liver fat content | Baseline measurement just prior to initiation of routine preoperative low calorie diet (this starts 3-4 weeks before surgery) compared to measurements on completion of this (within a week of surgery) and at 20% weight loss and 1 year after SG or RYGB
  Change in liver fat content as measured on MRI scan +/- fibroscan

SECONDARY OUTCOMES:
Hepatic fatty acid synthesis | liver biopsy taken during SG or RYGB
  measured by incorporation of 2H2 palmitate from 2H2O into very low density lipoprotein triglyceride (VLDL-TG) and contribution of de novo lipogenesis and uptake and re-esterification to the hepatic triglyceride pool in liver biopsy
Changes in relative contributions of pathways involved in lipid homeostasis | Baseline measurement just prior to initiation of routine preoperative low calorie diet (this starts 3-4 weeks before surgery) compared to measurements on completion of this (within a week of surgery) and at 20% weight loss and 1 year after SG or RYGB
  measured using mathematical modelling of results from stable isotope mixed meal test
Changes in fasting and postprandial plasma lipid concentration | Baseline measurements just prior to initiation of routine preoperative low calorie diet (this starts 3-4 weeks before surgery) compared to measurements on completion of this (within a week of surgery) and at 20% weight loss and 1 year after SG or RYGB
  measured using a clinical analyser (in fasting states and in response to mixed meal test)
Changes in fasting and postprandial plasma glucose concentration | Baseline measurement just prior to initiation of routine preoperative low calorie diet (this starts 3-4 weeks before surgery) compared to measurements on completion of this (within a week of surgery) and at 20% weight loss and 1 year after SG or RYGB
  measured using a clinical analyser measured using a clinical analyser (in fasting state and in response to mixed meal test)
Change in the incorporation of 13C (from dietary fat) into CO2 | Baseline measurement just prior to initiation of routine preoperative low calorie diet (this starts 3-4 weeks before surgery) compared to measurements on completion of this (within a week of surgery) and at 20% weight loss and 1 year after SG or RYGB
  measured using a breath analyser (in fasting state and in response to mixed meal test)
Expression changes (gene/protein) in adipose tissue biopsies | Baseline measurement just prior to initiation of routine preoperative low calorie diet (this starts 3-4 weeks before surgery) compared to measurements on completion of this (within a week of surgery) and at 20% weight loss and 1 year after SG or RYGB
  measured using techniques such as quantitative real-time PCR (polymerase chain reaction) and ELISA (enzyme- linked immunosorbent assay)
Change in fat mass | Baseline measurement just prior to initiation of routine preoperative low calorie diet (this starts 3-4 weeks before surgery) compared to measurements on completion of this (within a week of surgery) and at 20% weight loss and 1 year after SG or RYGB
  Proportional (% relative to baseline and lean mass) and absolute changes measured using DXA scan and bioimpedence analysis
Change in lean mass | Baseline measurement just prior to initiation of routine preoperative low calorie diet (this starts 3-4 weeks before surgery) compared to measurements on completion of this (within a week of surgery) and at 20% weight loss and 1 year after SG or RYGB
  Proportional (% relative to baseline and fat mass) and absolute changes measured using DXA scan and bioimpedence analysis
Change in functional strength | Baseline measurement just prior to initiation of routine preoperative low calorie diet (this starts 3-4 weeks before surgery) compared to measurements on completion of this (within a week of surgery) and at 20% weight loss and 1 year after SG or RYGB
  measured using hand dynamometer
changes in fasting and post-prandial peptides/proteins (e.g. PYY, GLP-1, insulin) | Baseline measurement just prior to initiation of routine preoperative low calorie diet (this starts 3-4 weeks before surgery) compared to measurements on completion of this (within a week of surgery) and at 20% weight loss and 1 year after SG or RYGB
  measured using ELISA (in fasting state and in response to mixed meal test)
change in weight | Baseline measurement just prior to initiation of routine preoperative low calorie diet (this starts 3-4 weeks before surgery) compared to measurements on completion of this (within a week of surgery) and at 20% weight loss and 1 year after SG or RYGB
  measured in kilograms using weighing scales
change in body mass index (BMI) | Baseline measurement just prior to initiation of routine preoperative low calorie diet (this starts 3-4 weeks before surgery) compared to measurements on completion of this (within a week of surgery) and at 20% weight loss and 1 year after SG or RYGB
  weight measured in kilograms using weighing scales and combined with height in metres to report BMI in kg/m^2
change in status of metabolic diseases (e.g. diabetes) / metabolic disease risk scores | Baseline measurement just prior to initiation of routine preoperative low calorie diet (this starts 3-4 weeks before surgery) compared to measurements on completion of this (within a week of surgery) and at 20% weight loss and 1 year after SG or RYGB
  measured with blood tests (e.g. hba1c), by recording clinical changes including medication requirements and clinical data (e.g. blood pressure)
complications, re-operation, mortality | Baseline measurement just prior to initiation of routine preoperative low calorie diet (this starts 3-4 weeks before surgery) compared to measurements on completion of this (within a week of surgery) and at 20% weight loss and 1 year after SG or RYGB
  clinical events will be recorded
changes in subcutaneous, visceral and pancreatic fat | Baseline measurement just prior to initiation of routine preoperative low calorie diet (this starts 3-4 weeks before surgery) compared to measurements on completion of this (within a week of surgery) and at 20% weight loss and 1 year after SG or RYGB
  measured on MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Tomlinson, MD PhD, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No